CLINICAL TRIAL: NCT04989842
Title: Studies on the Effectiveness and Equivalence of an Internet-based Virtual Classroom Intervention for Psychosomatic Aftercare According to the Hannover Curriculum
Brief Title: Effectiveness and Equivalence of an Internet-based Virtual Classroom Intervention for Psychosomatic Aftercare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Becker Hospital Group (Other)
Responsible Party: Principal Investigator, Dr. Alina Dahmen, Director, Dr. Becker Hospital Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Curriculum Hannover Online
Record Dates: First submitted 2021-07-14; First posted 2021-08-04 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Psychosomatic Disorder; Mental Disorder
Keywords: Rehabilitation; Psychosomatics; Aftercare; webbased aftercare therapy
MeSH Terms: conditions — Psychophysiologic Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group 1 (Active Comparator): webbased aftercare
  Interventions: Behavioral: Curriculum Hannover
- Control group (No Intervention): care as usual
- Intervention group 2 (Active Comparator): webbased aftercare
  Interventions: Behavioral: Curriculum Hannover
- face-to-face aftercare (Active Comparator): face-to-face aftercare
  Interventions: Behavioral: Curriculum Hannover

INTERVENTIONS:
Behavioral: Curriculum Hannover — The methodology uses a natural variation design within the Dr. Becker Clinical Group. The interventions consist of a face-to-face or a digital psychosomatic aftercare basing upon the concept of the Curriculum Hanover. A control group is included that does not receive these two interventions (but receives a similar rehabilitation treatment to the intervention groups).
  Arms: Intervention group 1; Intervention group 2; face-to-face aftercare

SUMMARY:
Outpatient psychosomatic aftercare after inpatient rehabilitation pursues the goal of helping patients to transfer the achieved rehabilitation result in everyday life and professional life. The Hanover Curriculum has been established as a treatment programme for psychosomatic aftercare. This comprises 25 weekly group sessions and two single therapies at the beginning and at the end of the therapy.

In Germany a vast majority of rehabilitants in a psychosomatic rehabilitation clinic has an indication for psychosomatic aftercare, but it is used only by less than half of the patients due to a lack of aftercare therapists. If there is a therapist in the patient's vicinity, there are often long travelling times to the therapist or the patients might feel stigmatized participating in a face-to-face therapy.

Thus, the expansion of internet-based aftercare services is recommended. Advantages are that they can be carried out at home, possible cost and time savings and improvement of the care situation.

Several meta-analyses provide high evidence for the effectiveness of internet-based therapy offers in depressive and anxiety disorders that are frequent among psychosomatic rehabilitation patients. First randomised controlled studies show that internet-based aftercare services can lead to a symptomatic improvement and to a reduction of relapses. It is currently not clear whether established aftercare concepts, such as the Curriculum Hannover, are also effective in an internet-based format (Curriculum Hannover Online).

The present project consists of a superiority study, examining whether participation in Curriculum- Hannover-Online leads to a stronger adoption and maintenance of the health improvements achieved in inpatient rehabilitation in comparison to care as usual, and an equivalnece study, examining, wether the Curriculum Hannover Online is an equivalent treatment option to the existing face-to-face aftercare therapy.

DETAILED DESCRIPTION:
The use of information and communication technology with the aim of promoting mental health can be described as "e-Mental Health", which is regularly used synonymously with the term "internet-based interventions".

With regard to the study situation on internet-based aftercare interventions, especially in Germany, the research is in an early phase. An overview of the possible uses of internet-based treatment approaches in rehabilitation can be found in Lin, Ebert, Lehr, Berking and Baumeister (2013) and - based on the contributions of the Rehabilitation Science Colloquium since 2008 - Baumeister, Lin and Ebert (2013). However, the first randomised controlled studies on aftercare show, in agreement with the studies outlined above, that corresponding offers led to a reduction in relapses compared to Care as Usual (CAU) (Bauer, Okon, Meermann, Kordy, 2013; Ebert, Tarnowski, Gollwitzer, Sieland& Berking, 2013).Both interventions represent new conceptual developments. Regarding the positive findings on the effectiveness of internet-based interventions and with a view to the suboptimal care situation, Kobelt, Winkler and Petermann (2011), for example, recommend the expansion of internet-based aftercare services and their evaluation.

The planned project aims to develop an internet-based variant of the aftercare concept Curriculum Hannover (Curriculum-Hannover-Online), to integrate it into routine care and to test its effectiveness. The technology of the virtual classroom is particularly suitable for internet-based interventions providing group therapy (cf. Wolever et al., 2012).

For this purpose, the existing manual for Curriculum Hannover (cf. Kobelt et al., 2002) is adapted in the course of the process for the needs of an online intervention. The therapists will be prepared for the specifics of the medium through a train-the-trainer-training for learning how to specifically establish and maintain a therapeutic relationship between therapist and participants. It is assumed that this new program for outpatient aftercare after inpatient psychosomatic rehabilitation can be an effective and useful therpy for patients who do not have access to the existing face-to-face aftercare therapies.. The Virtual Classroom is a direct, video- or audio-synchronous and multimedia contact between therapist and patient.

The main question of the superiority study is:

A. Does participation in the Curriculum-Hannover-Online lead to improved uptake and maintenance of the health improvements achieved in inpatient rehabilitation? B. Can the implementation of the Curriculum-Hannover-Online be designed in such a way that its use as a routine procedure in rehabilitation can be recommended? C. Can the Curriculum-Hannover-Online be accepted by the relevant stakeholders to the same extent as the face-to-face version of the Curriculum-Hannover-Online? For the successful introduction of a new treatment approach, in addition to the proof of its effectiveness, significant challenges have to be overcome with regard to the organisation of work processes, the involvement of all actors involved in the process (especially patients, practitioners, management).

The main question of the equivalence study is:

A.Does participation in the Curriculum-Hannover-Online lead to an equivalent adoption and maintenance of the health improvements achieved in inpatient rehabilitation? B. Can the implementation of the Curriculum-Hannover-Online in addition to the offer of the face-to-face variant be designed in such a way that its use as a rou- tine procedure in rehabilitation can be recommended? C.Can the Curriculum-Hannover-Online be accepted by the relevant stakeholders to the same extent as the face-to-face version of the Curriculum-Hannover-Online? D.Can characteristics be identified that allow a differential indication for the recommendation to participate in the Curriculum Hannover in its online or face-to-face variant? E.What are the additional advantages of the Curriculum Hannover Online from the perspective of patients, therapists, service providers and health care providers? Both studies will be conducted as two-arm randomised controlled trials. Individual rehabilitation patients will be randomised to the respective study arms. The system is based on a randomisation list (permuted blocks of variable length) with the help of the "Randlist" software at the sites. The order of the completed questionnaires determines the position in the list.

All data of the participants will be treated in accordance with the data security regulations (DSGVO), good scientific practice and the ethical requirements. Furthermore, all patients are informed about the project, ethics and data protection in a generally understandable way by a cover letter from their clinic before the treatment. All project staff are obliged to comply with the ethics guidelines and to maintain confidentiality. The pre- and post-data of the patients are combined by means of a personal code, which does not allow any conclusion about the participant.

ELIGIBILITY:
Inclusion Criteria:

* Patients after psychosomatic rehabilitation
* indication for outpatient psychosomatic aftercare are included in both studies.
* access to a standard PC and broadband internet connection is required (DSL or LTE).

Exclusion Criteria:

Persons who are

* are discharged with a capacity of less than three hours per day on the general labour market,
* receive or have applied for a pension of at least two-thirds of the full pension,
* receive a benefit that is regularly paid until the start of an old-age pension.
* suffering from acute addiction disorder / acute psychosis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6023 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
change of psychic and somatoform complaints | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)

SECONDARY OUTCOMES:
change of depressiveness | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of phobic anxiety | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of somatoform complaints | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of mental well-being | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of interactional difficulties | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of self-efficacy | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of activity and participation | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of social support | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of social stress | up to 18 months
  according to the HEALTH-49 (Rabung et al., 2009)
change of employment prognosis | up to 18 months
  according to the subjective employment forecast (Mittag et al.,2006)
change of workability | up to 18 months
  according to the work ability index (Hasselhorn&Freude, 2007)

CONTACTS AND LOCATIONS:
Overall Officials: Alina Dahmen, MD, Study Director — Dr. Becker Hospital Group
Locations (1):
- Dr. Becker Hospital Group, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be published. Other researchers are welcome to get in contact with the PI to get access to anonymous data.

REFERENCES:
- [Background] Andersson G, Cuijpers P, Carlbring P, Riper H, Hedman E. Guided Internet-based vs. face-to-face cognitive behavior therapy for psychiatric and somatic disorders: a systematic review and meta-analysis. World Psychiatry. 2014 Oct;13(3):288-95. doi: 10.1002/wps.20151. PMID 25273302
- [Background] Arnberg FK, Linton SJ, Hultcrantz M, Heintz E, Jonsson U. Internet-delivered psychological treatments for mood and anxiety disorders: a systematic review of their efficacy, safety, and cost-effectiveness. PLoS One. 2014 May 20;9(5):e98118. doi: 10.1371/journal.pone.0098118. eCollection 2014. PMID 24844847
- [Background] Cheng SK, Dizon J. Computerised cognitive behavioural therapy for insomnia: a systematic review and meta-analysis. Psychother Psychosom. 2012;81(4):206-16. doi: 10.1159/000335379. Epub 2012 May 11. PMID 22585048
- [Background] Cuijpers P, van Straten A, Warmerdam L, van Rooy MJ. Recruiting participants for interventions to prevent the onset of depressive disorders: possible ways to increase participation rates. BMC Health Serv Res. 2010 Jun 25;10:181. doi: 10.1186/1472-6963-10-181. PMID 20579332
- [Background] Cuijpers P, Marks IM, van Straten A, Cavanagh K, Gega L, Andersson G. Computer-aided psychotherapy for anxiety disorders: a meta-analytic review. Cogn Behav Ther. 2009;38(2):66-82. doi: 10.1080/16506070802694776. PMID 20183688
- [Background] Ebert DD, Lehr D, Boss L, Riper H, Cuijpers P, Andersson G, Thiart H, Heber E, Berking M. Efficacy of an internet-based problem-solving training for teachers: results of a randomized controlled trial. Scand J Work Environ Health. 2014 Nov;40(6):582-96. doi: 10.5271/sjweh.3449. Epub 2014 Aug 13. PMID 25121986
- [Background] Ebert D, Tarnowski T, Gollwitzer M, Sieland B, Berking M. A transdiagnostic internet-based maintenance treatment enhances the stability of outcome after inpatient cognitive behavioral therapy: a randomized controlled trial. Psychother Psychosom. 2013;82(4):246-56. doi: 10.1159/000345967. Epub 2013 Jun 1. PMID 23736751
- [Background] Haug T, Nordgreen T, Ost LG, Havik OE. Self-help treatment of anxiety disorders: a meta-analysis and meta-regression of effects and potential moderators. Clin Psychol Rev. 2012 Jul;32(5):425-45. doi: 10.1016/j.cpr.2012.04.002. Epub 2012 Apr 21. PMID 22681915
- [Background] Lin J, Ebert DD, Lehr D, Berking M, Baumeister H. [Internet based cognitive behavioral interventions: state of the art and implementation possibilities in rehabilitation]. Rehabilitation (Stuttg). 2013 Jun;52(3):155-63. doi: 10.1055/s-0033-1343491. Epub 2013 Jun 12. German. PMID 23761204
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. BMJ. 2010 Mar 23;340:c869. doi: 10.1136/bmj.c869. No abstract available. PMID 20332511
- [Background] Wolever RQ, Bobinet KJ, McCabe K, Mackenzie ER, Fekete E, Kusnick CA, Baime M. Effective and viable mind-body stress reduction in the workplace: a randomized controlled trial. J Occup Health Psychol. 2012 Apr;17(2):246-258. doi: 10.1037/a0027278. Epub 2012 Feb 20. PMID 22352291
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Derived] Lippke S, Gao L, Keller FM, Becker P, Dahmen A. Adherence With Online Therapy vs Face-to-Face Therapy and With Online Therapy vs Care as Usual: Secondary Analysis of Two Randomized Controlled Trials. J Med Internet Res. 2021 Nov 3;23(11):e31274. doi: 10.2196/31274. PMID 34730541